CLINICAL TRIAL: NCT00210613
Title: A Placebo-Controlled, Double-Blind, Randomized, Parallel Study of the Withdrawal Effects of Chronic Daily and As-Needed Dosing With Dapoxetine in the Treatment of Premature Ejaculation
Brief Title: A Study of Withdrawal Effects With Dapoxetine in the Treatment of Premature Ejaculation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003451
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-12

CONDITIONS: Sexual Dysfunction; Ejaculation
Keywords: dapoxetine; premature ejaculation; sexual dysfunction; orgasmic disorder; sexual intercourse; ejaculation
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Premature Ejaculation; Sexual Dysfunctions, Psychological; Coitus | interventions — dapoxetine

INTERVENTIONS:
Drug: Dapoxetine

SUMMARY:
The primary purpose of the study is to assess the possible withdrawal effects after abruptly stopping daily therapy with dapoxetine compared with continuing daily therapy in men with premature ejaculation (PE).

DETAILED DESCRIPTION:
Premature ejaculation (PE) is a form of male sexual dysfunction. A measure of withdrawal effects associated with stopping therapy for PE is the Discontinuation-Emergent Signs and Symptoms (DESS), a series of questions for signs and symptoms experienced by the patient. This study of men with PE is a multicenter, randomized, double-blind trial consisting of 3 phases: pre-randomization phase (a screening visit and 1-week baseline period); 10-week double-blind treatment phase during which patients receive dapoxetine or placebo; and 2-week follow-up phase. The total duration of the study is approximately 13 weeks. During the double-blind phase patients receive study medication for once daily treatment and for use on as "as-needed" basis prior to sexual activity. After 9 weeks, some patients (half of the active patients) continue treatment with dapoxetine and other (another half of the active patients) are switched to placebo for the last week of therapy, abruptly stopping the study drug. Assessments of effectiveness include the incidence of withdrawal symptoms, assessed by changes in DESS; control over ejaculation, satisfaction with sexual intercourse, and severity of symptom impressions, based on questions asked at specified intervals during the study. Safety assessments include the incidence, severity, and type of adverse events throughout the study, as well as laboratory tests and questionnaires to monitor sexual function at specified times during the study.The study hypothesis is that abruptly stopping treatment with dapoxetine in men with PE does not result in an increase in withdrawal symptoms (as assessed by DESS), compared with the men who stay with the treatment. Oral tablets of dapoxetine (60 milligrams) taken once daily and also as needed during 10 weeks of treatment. No more than 1 tablet for daily treatment and 1 as-needed tablet within a 24-hour period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is in a stable, monogamous sexual relationship with the same woman for at least 6 months and plans to maintain this relationship for the duration of the study
* diagnosis of premature ejaculation (PE) according to the criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) for at least 6 months before study initiation
* experience PE in the majority of sexual intercourse events
* good general health at study initiation
* patient and partner willing to avoid situations or activities that may have an effect o their sexual activity (for example, avoid pregnancy, refrain from any preplanned surgery)

Exclusion Criteria:

* Not taken dapoxetine or participated in another study investigating pharmacologic treatment of PE within the last 3 months
* no history of any medical events such as surgery, injury, infections, or neurological conditions that are associated with the development of PE
* not taken an investigational drug within 1 month, or used an experimental medical device within 6 months, of study initiation
* no positive diagnosis of depressive or anxiety disorder, manic episode, panic disorder, obsessive-compulsive disorder, posttraumatic stress disorder, alcohol abuse and dependence, schizophrenia, or other psychotic disorders
* no known allergy or hypersensitivity to selective serotonin reuptake inhibitors (SSRIs) or serotonin norepinephrine reuptake inhibitors (SNRIs)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2004-11; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Incidence of withdrawal symptoms (defined by a checklist of signs and symptoms associated with stopping the therapy) at Weeks 9, 10, and 11 of treatment

SECONDARY OUTCOMES:
Control over ejaculation, satisfaction with sexual intercourse, and severity of symptom impressions, based on questions asked at start of study through Week 11; adverse incidence and severity throughout study and follow up (Week 12)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Background] Porst H, McMahon CG, Althof SE, Sharlip I, Bull S, Aquilina JW, Tesfaye F, Rivas DA. Baseline characteristics and treatment outcomes for men with acquired or lifelong premature ejaculation with mild or no erectile dysfunction: integrated analyses of two phase 3 dapoxetine trials. J Sex Med. 2010 Jun;7(6):2231-2242. doi: 10.1111/j.1743-6109.2010.01820.x. Epub 2010 Apr 19. PMID 20412423
- [Derived] McMahon CG, Althof SE, Kaufman JM, Buvat J, Levine SB, Aquilina JW, Tesfaye F, Rothman M, Rivas DA, Porst H. Efficacy and safety of dapoxetine for the treatment of premature ejaculation: integrated analysis of results from five phase 3 trials. J Sex Med. 2011 Feb;8(2):524-39. doi: 10.1111/j.1743-6109.2010.02097.x. Epub 2010 Nov 8. PMID 21059176
- See also: A Placebo-Controlled, Double-Blind, Randomized, Parallel Study of the Withdrawal Effects of Chronic Daily and As-Needed Dosing With Dapoxetine in the Treatment of Premature Ejaculation. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=529&filename=CR003451_CSR.pdf